CLINICAL TRIAL: NCT01253668
Title: Brivanib (BMS-582664, Brivanib Alaninate) in Treatment of Refractory Metastatic Renal Cell Carcinoma - A Phase II Pharmacodynamic and Baseline Biomarker Study
Brief Title: Brivanib Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: In November 2012, this study was permanently closed to new accrual at the request of the drug manufacturer (BMS), who decided not to pursue additional research activity in this patient population.
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 04810
Record Dates: First submitted 2010-11-30; First posted 2010-12-03 (Estimated); Results first posted 2021-03-19 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — brivanib; Polymerase Chain Reaction; Magnetic Resonance Spectroscopy; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Patients receive oral brivanib alaninate daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brivanib alaninate; Genetic: Polymerase chain reaction; Other: Iodine I 124 chimeric monoclonal antibody G250; Procedure: Positron emission tomography/computed tomography; Genetic: Protein expression analysis; Other: Immunohistochemistry

INTERVENTIONS:
Drug: Brivanib alaninate — Brivanib by mouth daily at a dose of 800mg.
Genetic: Polymerase chain reaction — Undergo 1241-cG250 PET/CT imaging (correlative studies)
  Other Names: PCR
Other: Iodine I 124 chimeric monoclonal antibody G250 — Undergo 124I-cG250 PET/CT imaging (correlative studies)
Procedure: Positron emission tomography/computed tomography — Undergo 1241-cG250 PET/CT imaging (correlative studies)
Genetic: Protein expression analysis — Correlative studies
Other: Immunohistochemistry — correlative studies
  Other Names: immunohistochemistry staining method

SUMMARY:
This is a phase II study of an investigational agent, brivanib, in patients with refractory metastatic renal cell carcinoma. This study will evaluate the safety and effectiveness of brivanib in renal cell carcinoma, and explore the activity of this drug in this population to determine whether imaging and molecular features of the tumors can be used to predict response. Approximately 30 people with advanced kidney cancer will be enrolled on this study at the University of Pennsylvania.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to determine the efficacy of brivanib in the treatment of metastatic renal cell carcinoma in terms of progression-free survival (PFS) in patients who have progressed on treatment with sunitinib, sorafenib, bevacizumab, or pazopanib. The primary endpoint of the trial will be PFS at 16 weeks. The secondary objectives are to further examine the safety and tolerability profile of brivanib, to examine the efficacy of brivanib in this population in terms of best overall response, response rate, progression-free survival, and overall survival, to describe baseline and changes in I-cG250 PET/CT in relation to observed therapeutic effects, to describe novel baseline histologic features of these tumors in relation to observed therapeutic effects. Modalities will include Von Hippel-Lindau gene (VHL) and hypoxia-inducible factor 1 gene (HIF-1) expression assessment and a novel histo-cytometric assessment of the tumor microenvironment in terms of p-STAT3, p-ERK, Ki67, VEGFR2, FGFR1 expression, to describe changes in circulating collagen IV on brivanib in relation to therapeutic effects, to explore the relationship between single nucleotide polymorphisms in angiogenesis-related genes and the activity of brivanib in the treatment of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults with metastatic renal cell carcinoma
* Patients will have tumors that bear a clear cell component that comprises greater than or equal to 50% of the tumor.
* Disease must be measurable in accord with RECIST 1.1 guidelines.
* Patients who have developed progressive disease or intolerance on treatment with sorafenib, sunitinib, bevacizumab, or pazopanib over a 60 day period who have not discontinued this therapy more than 100 days prior to study enrollment. Progressive disease per RECIST 1.1 guidelines will be preferred
* Therapy with up to three prior systemic regimens will be allowed.
* Patients may have been treated with any of the following: sorafenib, sunitinib, bevacizumab, pazopanib, temsirolimus, everolimus, interferon alpha, interleuken-2.
* Treatment with up to one prior regimen that included cytotoxic chemotherapy will be allowed.
* Patients may have been treated with more than 1 antiangiogenic therapy (e.g., patients may have been treated with both sorafenib and sunitinib or sunitinib and bevacizumab, or sequential combinations that include pazopanib).
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Tumor tissue must be available for correlative studies.
* Patients must consent to allow the acquisition of formalin-fixed paraffin-embedded (FFPE) material (block or unstained slides) by study personnel for performance of correlative tissue studies.

Exclusion Criteria:

* Known brain metastases
* Prior therapy with brivanib, or anti-FGFR (fibroblast growth factor receptor) therapy.
* History of thrombotic or embolic events within the last six months such as a cerebrovascular accident (including transient ischemic attacks), pulmonary embolism.
* Gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE version 4.0 Grade greater than 3 within 30 days prior to study entry.
* Uncontrolled or significant cardiovascular disease.
* QTc greater than 450 msec on two consecutive ECGs (Baseline ECG should be repeated if QTc is found to be greater than 450 msec.).
* Active infection, less than 7 days after completing systemic antibiotic therapy.
* History of non-healing wounds or ulcers or bone fractures within 3 months of fracture.
* Major surgical procedure, open biopsy, or significant traumatic injury less than 3 weeks prior to study enrollment or those who receive minor surgical procedures (e.g. core biopsy or fine needle aspiration)within 1 week prior to study enrollment.
* Cytotoxic chemotherapy within 3 weeks, bevacizumab within 2 months, or radiation therapy within 2 weeks, other targeted therapies (e.g., sorafenib, sunitinib, temsirolimus, everolimus)within 2 days.
* Inability to swallow tablets or untreated malabsorption syndrome.
* Pre-existing thyroid abnormality with thyroid function that cannot be controlled with medication.
* History of HIV
* Patients with centrally cavitating lung lesions.
* Patients requiring therapeutic anticoagulation with warfarin at baseline. However, prophylactic therapy with a low molecular weight heparin at baseline is acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Keefe, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1
Started (The study was terminated, and the PI has left the institution. Despite all possible efforts to contact the PI/study team members, no data are available to be reported.) | 0
Completed (The study was terminated, and the PI has left the institution. Despite all possible efforts to contact the PI/study team members, no data are available to be reported) | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated, and the PI has left the institution. Despite all possible efforts to contact the PI/study team members, no data are available to be reported
Arm/Group | Arm 1
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: All patients will be followed through the entire 16-week period and will be given a binary outcome assignment: progressive disease or not.
Time Frame: 16 weeks
Population: as for baseline characteristics
Arm/Group | Arm 1
Number analyzed (Participants) | 0

2. Secondary Outcome: Best Overall Response Rated for Each Patients as Assessed by RECIST 1.1 Guidelines
Description: The best overall radiographic response to therapy as measured and assessed using RECIST 1.1 guidelines will be captured for each research subject.
Time Frame: Every 8 weeks
Population: as for baseline characteristics
Arm/Group | Arm 1
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Will record deaths on study, and, to the extent possible, after the study follow-up period is completed for each patient, will be captured. Reason for death will be identified and recorded where possible.
Time Frame: Every 8 weeks
Population: as for baseline characteristics
Arm/Group | Arm 1
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Total Antibody Binding as Assessed by 124I-cG250 PET/CT Imaging (Correlative Studies)
Description: Will determine the baseline and change in total antibody binding in lesions from baseline to the time on treatment that patients are assessed. The analysis dataset will be quantitated radiotracer uptake data obtained via I-cG250 PET/CT for all evaluable patients who complete the trial.
Time Frame: At baseline and 8 weeks
Population: as for baseline characteristics
Arm/Group | Arm 1
Number analyzed (Participants) | 0

5. Secondary Outcome: Response Rate for All Patients
Description: Response Rate for all patients as assessed by RECIST 1.1 guidelines
Time Frame: Every 8 weeks
Population: as for baseline characteristics
Arm/Group | Arm 1
Number analyzed (Participants) | 0

6. Secondary Outcome: Molecular Markers
Description: Molecular markers expressed in patient tumor specimens as assessed by IHC and histocytometry (e.g., VHL, HIF, p-STAT3, p-ERK, and Ki67, VEGFR2, and FGFR1) (correlative studies)
Time Frame: At baseline
Population: as for baseline characteristics
Arm/Group | Arm 1
Number analyzed (Participants) | 0

7. Secondary Outcome: Changes in Collagen IV Levels
Description: Changes in collagen IV levels for each patient (correlative studies)
Time Frame: At baseline and week 3
Population: as for baseline characteristics
Arm/Group | Arm 1
Number analyzed (Participants) | 0

8. Secondary Outcome: Germline Polymorphisms and Assessment of Relationship to Toxicity and Clinical Outcome
Description: Germline polymorphisms and assessment of relationship to toxicity and clinical outcome (correlative studies)
Time Frame: At baseline and week 3
Population: as for baseline characteristics
Arm/Group | Arm 1
Number analyzed (Participants) | 0

9. Secondary Outcome: Blood Pressure Data
Description: Blood pressure data
Time Frame: At baseline, day 1 weeks 3,6,8,12,16 and every 6-8 weeks thereafter
Population: as for baseline characteristics
Arm/Group | Arm 1
Number analyzed (Participants) | 0

10. Secondary Outcome: Toxicity as Assessed by NCI CTCAE Version 4.0
Description: Toxicity as assessed by NCI CTCAE version 4.0
Time Frame: Day 1, weeks 3,6,9,12,16, and every 6-8 weeks thereafter
Population: as for baseline characteristics
Arm/Group | Arm 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The study was terminated, and the PI has left the institution. Despite all possible efforts to contact the PI/study team members, no data are available to be reported.
Description: The study was terminated, and the PI has left the institution. Despite all possible efforts to contact the PI/study team members, no data are available to be reported.
Arm/Group | Arm 1
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated, and the PI has left the institution. Despite all possible efforts to contact the PI/study team members, no data are available to be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No